CLINICAL TRIAL: NCT00006078
Title: Single Dose Pharmacokinetic Study of Lycopene Delivered in a Well Defined Food-Based Lycopene Delivery System (Tomato Paste-oil Mixture) in Healthy Male Volunteers Between 18 and 45 Years of Age
Brief Title: Lycopene In Preventing of Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Prevention
Other Study IDs: UIC-H-99-058; CDR0000067915 (Registry Identifier: PDQ (Physician Data Query)); UIC-N01-CN-85081; NCI-P00-0143
Record Dates: First submitted 2000-08-03; First posted 2003-01-27 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2004-12

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lycopene

INTERVENTIONS:
Dietary Supplement: lycopene

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development of cancer. The use of lycopene may be an effective way to prevent prostate cancer.

PURPOSE: Phase I trial to study the effectiveness of lycopene in preventing prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine any dose limiting toxicities and the maximum tolerated dose of lycopene administered orally as a food based delivery system in healthy male subjects 18-45 years of age for the chemoprevention of prostate cancer.
* Determine the pharmacokinetics of this regimen in this population.
* Determine the dose range of this regimen to be used in the 3 month multiple dose study, based on the toxicity, pharmacokinetics and feasibility resulting from the present study in this population.

OUTLINE: This is a dose-escalation study.

Patients receive a single dose of oral lycopene in a mixture of tomato paste, water, and olive oil over 15 minutes on day 1. Patients are asked to maintain a diet that contains negligible carotinoid for 28 days.

Cohorts of 5 patients receive escalating doses of lycopene until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 5 patients experience dose limiting toxicities.

Patients are followed weekly for 4 weeks.

PROJECTED ACCRUAL: A total of 5-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Normal healthy males judged to be in good medical condition based on history and physical exam confirming the absence of chronic medical conditions
* Baseline serum lycopene less than 600 nM

PATIENT CHARACTERISTICS:

Age:

* 18 to 45

Performance status:

* Karnofsky 100%

Life expectancy:

* Not specified

Hematopoietic:

* Hematologic function normal

Hepatic:

* Liver function normal
* No hepatic disease

Renal:

* Kidney function normal
* No renal disease

Cardiovascular:

* No hypertension requiring medication
* No cardiovascular disease
* Normal EKG

Other:

* No evidence of a psychiatric disorder
* Must be within 15% of ideal body weight based on standard weight tables
* No history of smoking within the past 3 months
* At least 72 hours since prior alcohol consumption and no history of alcohol abuse
* No history of gastrointestinal malabsorption or any other condition that could affect drug absorption
* No allergy to tomato based products
* No active malignancy at any site
* No illness that would pose a threat or additional risk (e.g., thyroid disease, diabetes mellitus)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* At least 14 days since prior prescription drugs
* No concurrent regular prescription medications
* At least 30 days since other prior experimental drugs
* No concurrent participation in any other experimental trial

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2000-06; Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith A. Rodvold, Study Chair — University of Illinois at Chicago
Locations (1):
- University of Illinois Medical Center, Chicago, Illinois, United States